CLINICAL TRIAL: NCT01130805
Title: A Phase II Study of Pazopanib in Combination With Capecitabine and Oxaliplatin (CAPEOX) in Patients With Advanced Gastric Cancer
Brief Title: A Study of Pazopanib With CAPEOX in AGC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joon Oh Park, associate professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-03-068
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Gastric Cancer
Keywords: gastric cancer pazopanib capecitabine, oxaliplatin; Metastatic or recurrent gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — pazopanib; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib in combination with capecitabine and oxaliplatin (Experimental): Capecitabine 850 mg/m2 bid on day 1-14, Oxaliplatin 130 mg/m2 IV on day 1 and Pazopanib 800 mg once in a day on day 1-21, every 3 weeks
  Interventions: Drug: Pazopanib in combination with capecitabine and oxaliplatin

INTERVENTIONS:
Drug: Pazopanib in combination with capecitabine and oxaliplatin — Capecitabine 850 mg/m2 bid on day 1-14, Oxaliplatin 130 mg/m2 IV on day 1 and Pazopanib 800 mg once in a day on day 1-21, every 3 weeks
  Other Names: Capecitabine, Oxaliplatin, pazopanib

SUMMARY:
In order to improve survival of metastatic gastric cancer patients, we plan to to conduct a phase II trial of CapeOx with 800 mg once-daily pazopanib as a first-line chemotherapy in metastatic gastric cancer patients.

DETAILED DESCRIPTION:
Despite improvements in the early diagnosis of gastric cancer, many patients present with inoperable disease and an effective, novel combination treatment is urgently needed for these patients population. A recent meta-analysis demonstrated that chemotherapy improves survival for patients with advanced gastric cancer compared with best supportive care alone [hazard ratio (HR) 0.39, 95% confidence interval (CI) 0.28-0.52] and that combination chemotherapy is superior to monotherapy (HR 0.83, 95% CI 0.74-0.93) (Wagner et al., 2006). For advanced gastric cancer, 5-FU in combination with cisplatin (FP regimen) is commonly used reference regimen, which are successfully replaced by capecitabine and oxaliplatin in recent phase III trial (Cunningham et al., 2008; Okines et al., 2009). In phase II trial, CAPEOX (capecitabine combined with oxaliplatin) regimen also showed promising activity for the metastatic gastric cancer (Park et al., 2006; Park et al., 2008). In order to improve survival of metastatic gastric cancer patients, various clinical trials incorporated novel molecularly targeted agent in combination with the reference arm.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who provide written informed consent
* Age over 18 years
* Histologically proven unresectable gastric cancer
* ECOG performance status of 0-2
* At least one uni-dimensionally measurable lesion by RECIST criteria ver 1.1
* Adequate organ system function absolute neutrophil count > 1,500/µL, platelets > 100,000/µL, hemoglobin > 9g/dl Total bilirubin < 1.5 times upper limit of normal (ULN), AST and ALT < 2.5 times ULN, PT (INR), PTT < 1.2 times UNL Serum creatinine less than 1.5 mg/dL or Calculated Ccr at least 50 mL/min, Urine Protein to Creatinine Ratio (UPC) less than 1
* female with Non-childbearing potential

Exclusion Criteria:

* Prior malignancy
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product
* Presence of uncontrolled infection
* Corrected QT interval (QTc) above 480 msecs using Bazett's formula
* History of any one or more of the following cardiovascular conditions within the past 6 months: Cardiac angioplasty or stenting, Myocardial infarction, Unstable angina, Coronary artery bypass graft surgery, Symptomatic peripheral vascular disease, Class II or higher congestive heart failure
* Poorly controlled hypertension while on antihypertensive agents
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer
* Evidence of active bleeding or bleeding diathesis
* Hemoptysis within 6 weeks of first dose of study drug
* Any serious and/or unstable preexisting medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Unable or unwilling to discontinue use of prohibited medications listed in the protocol
* Treatment with any of the following anti-cancer therapies;Radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib; biologic therapy, immunotherapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib; No prior chemotherapy except adjuvant chemotherapy (Patients who received adjuvant chemotherapy at least 6 months prior to study entry will be allowed regardless of chemotherapeutic regimen
* Pre-existing grade 2 (or higher) motor or sensory neuropathy by CTCAE v4.0
* Known allergy to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-12; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 months after last patient

SECONDARY OUTCOMES:
Progression free survival (PFS) | one year
Overall survival (OS) | Two years
Metabolic response rate by PET-CT | 1 month
Toxicities | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joon Oh Park, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Kim ST, Lee J, Lee SJ, Park SH, Jung SH, Park YS, Lim HY, Kang WK, Park JO. Prospective phase II trial of pazopanib plus CapeOX (capecitabine and oxaliplatin) in previously untreated patients with advanced gastric cancer. Oncotarget. 2016 Apr 26;7(17):24088-96. doi: 10.18632/oncotarget.8175. PMID 27003363
- [Derived] Kim ST, Ahn S, Lee J, Lee SJ, Park SH, Park YS, Lim HY, Kang WK, Kim KM, Park JO. Value of FGFR2 expression for advanced gastric cancer patients receiving pazopanib plus CapeOX (capecitabine and oxaliplatin). J Cancer Res Clin Oncol. 2016 Jun;142(6):1231-7. doi: 10.1007/s00432-016-2143-2. Epub 2016 Mar 16. PMID 26983912